CLINICAL TRIAL: NCT01996800
Title: The Effects of Spinal Manipulative Therapy and Neuromuscular Reeducation on the Presentation of Autistic Symptoms in Children
Brief Title: Study of Chiropractic and Neuromuscular Reeducation as a Treatment for Autism Symptoms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient faculty and staff.
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SCU-AUT-01
Record Dates: First submitted 2013-11-05; First posted 2013-11-27 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Manipulative Therapy (SMT) (Experimental): Patients will receive 12 weeks of chiropractic SMT
  Interventions: Procedure: Spinal Manipulative Therapy (SMT)
- SMT and Neuromuscular Reeducation (Active Comparator): Spinal manipulation is a therapeutic intervention performed on spinal articulations which are synovial joints. These articulations in the spine that are amenable to spinal manipulative therapy include the z-joints, the atlanto-occipital, atlanto-axial, lumbosacral, sacroiliac, costotransverse and costovertebral joints.
  A neuromuscular re-education program will consist of repetitive movements, posturing, and stimulation designed to reinforce nerve signals for functional movements. It is theorized that when the nerve signals are "retrained" and appropriate muscle movements are repeated, movement patterns become automatic again. Neuromuscular re-education is usually done along with other types of treatment to promote functional muscle movement.
  Interventions: Procedure: Spinal Manipulative Therapy (SMT); Procedure: SMT and Neuromuscular Reeducation

INTERVENTIONS:
Procedure: Spinal Manipulative Therapy (SMT) — Spinal manipulation is a therapeutic intervention performed on spinal articulations which are synovial joints. These articulations in the spine that are amenable to spinal manipulative therapy include the z-joints, the atlanto-occipital, atlanto-axial, lumbosacral, sacroiliac, costotransverse and costovertebral joints.
Procedure: SMT and Neuromuscular Reeducation — Neuromuscular reeducation is a general term that refers to techniques that attempt to retrain the neuromuscular system to function properly. The basis of this idea is that the formation of certain patterns of communication between muscles and nerves allow people to perform simple everyday acts such as climbing stairs.
  Arms: SMT and Neuromuscular Reeducation

SUMMARY:
This study explores the effectiveness of chiropractic and neuromuscular reeducation as complementary and alternative medicine treatment approaches for autism. Our investigation maintains the following three hypotheses:

1. Spinal manipulative therapy (SMT) will reduce the presentation of autistic symptoms in children.
2. Spinal manipulative therapy (SMT) in conjunction with neuromuscular reeducation will reduce the presentation of autistic symptoms in children.
3. The presentation of autistic symptoms in children will significantly differ between the treatment groups of spinal manipulative therapy and spinal manipulative therapy in unification with neuromuscular reeducation.

DETAILED DESCRIPTION:
We aim to describe and illustrate the roles of spinal manipulative therapy and neuromuscular reeducation in autistic children at a CAM university health center with regard to the following:

1. To measure the safety and efficacy of spinal manipulative therapy for the autism spectrum disorders
2. To measure the safety and efficacy of spinal manipulative therapy and neuromuscular reeducation for the treatment of the autism spectrum disorders
3. To begin to establish or debunk debated SMT treatment for autism
4. To evaluate, gauge, and improve current autism assessment tools by exploring face validity of the measures as indicated by ongoing data collection

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed by a physician with an Autism Spectrum Disorder between the ages of 5 and 15
* Children with parents able to bring their child to the university health center two times a week for 12 weeks
* Children assessed to have a level of functioning that is conducive to experiencing and undergoing chiropractic treatment at the university health center.
* Children without the presentation and diagnosis of comorbidity

Exclusion Criteria:

* Children with comorbidity or multiple diagnoses (mental retardation, chromosomal disorders)
* Children undergoing another treatment for their disorder, other than a form of behavioral therapy (ABA or DTT) by a trained or licensed mental health professional.
* Children taking medication that is not deemed to be stabilized by a primary care physician, including medication dosages that is likely to be shifted and changed during the 12 weeks of treatment in this investigation.
* Children assessed to have severe behavioral impediments not conducive to chiropractic treatment at the university health center.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessing change using the Autism Treatment Evaluation Checklist | Weeks 1, 6, and 12
  Please see:
  Rimland, B., & Edelson, S. M. (2000). Autism treatment evaluation checklist (ATEC). Retrieved October, 23, 2006.
  Volkmar, F. R., Cicchetti, D. V., Dykens, E., Sparrow, S. S., Leckman, J. F., & Cohen, D. J. (1988). An evaluation of the autism behavior checklist. Journal of Autism and Developmental Disorders, 18(1), 81-97.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Korgan, PhD, Principal Investigator — Southern California University of Health Sciences; Rochelle Neally, DC, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: No